CLINICAL TRIAL: NCT00005716
Title: Asthma Partnership for Minority Children
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4925; R01HL052833 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2002-05

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To evaluate the efficacy of a community-based intervention to improve asthma management for parents, children and health care providers.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Forty-two (42) elementary schools in urban Baltimore and Washington, DC, served as recruitment sites and approximately 300 students with moderate to severe asthma were enrolled. All participants enrolled in the A+ Asthma Program. Primary care practitioners of these students were randomized to a minimal contact program or to the A+ asthma physician partnership. They were offered a menu of educational offerings to improve their knowledge and skills. The primary outcome measure was emergency care use. Secondary measures included physician practices, hospitalization, health care utilization, restricted activities, medication use, school absences and coping skills.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-08; Study Completion 1999-07 (Actual)

REFERENCES:
- [Background] Allen FC, Vargas PA, Kolodner K, Eggleston P, Butz A, Huss K, Malveaux F, Rand CS. Assessing pediatric clinical asthma practices and perceptions: a new instrument. J Asthma. 2000 Feb;37(1):31-42. doi: 10.3109/02770900009055426. PMID 10724296
- [Background] Butz AM, Eggleston P, Huss K, Kolodner K, Rand C. Nebulizer use in inner-city children with asthma: morbidity, medication use, and asthma management practices. Arch Pediatr Adolesc Med. 2000 Oct;154(10):984-90. doi: 10.1001/archpedi.154.10.984. PMID 11030849
- [Background] Bartlett SJ, Kolodner K, Butz AM, Eggleston P, Malveaux FJ, Rand CS. Maternal depressive symptoms and emergency department use among inner-city children with asthma. Arch Pediatr Adolesc Med. 2001 Mar;155(3):347-53. doi: 10.1001/archpedi.155.3.347. PMID 11231800